CLINICAL TRIAL: NCT05020639
Title: A Phase I Study to Evaluate the Tolerability and Pharmacokinetics of TQB3820 in Relapsed or Refractory Multiple Myeloma (R/R MM) or Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma (R/R B-NHL)
Brief Title: A Study of TQB3820 in Patients With Hematological Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3820-I-01
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3820 tablets (Experimental): TQB3820 tablets are administrated orally on Days 1-28 of each 28-day treatment cycle. Dose escalation of TQB3820 will be based on evaluation of clinical safety and tolerability and guided by accumulating PK data.
  Interventions: Drug: TQB3820 tablets

INTERVENTIONS:
Drug: TQB3820 tablets — TQB3820 is a novel cereblon-modulating agent.

SUMMARY:
TQB3820 is a novel cereblon-modulating agent. Upon binding to cereblon, a substrate receptor in the cullin4 E3 ligase complex, TQB3820 promotes recruitment, ubiquitination, and subsequent proteasomal degradation of the hematopoietic transcription factors Ikaros (IKZF1) and Aiolos (IKZF3). Modulation of Aiolos and Ikaros expression has the potential to correct multiple aspects of the immune dysregulation mediated by B cells.

ELIGIBILITY:
Inclusion Criteria:

1. For Multiple Myeloma cohort

   1. Patients must have received at least 2 prior therapies;
   2. Measurable levels of myeloma paraprotein

      1. M-protein in serum >5 g/L;
      2. M-protein in urine >200mg/24h;
      3. Light chain Multiple Myeloma without measurable disease in the serum or urine: serum immunoglobulin free light chain ≥ 100 mg/L and abnormal serum immunoglobulin kappa lambda free light chain ratio.
2. For Indolent B-NHL

   1. Progressed after standard treatment or no standard treatment with an established survival benefit is available;
   2. Imaging in screening showing at least one measurable lesion; In patients with CLL/SLL, circulating lymphocytes >= 5.0 × 10^9/L or lesions greater than 1.5 cm.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
4. Life expectancy >=3 months;
5. Adequate organ/system function;
6. Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped;

Exclusion Criteria:

1. Patients received allogenic haemopoietic stem cell transplantation, or autologous stem cell transplantation within 3 months;
2. Diagnosed and/or treated additional malignancy within 3 years before the first dose;
3. With factors affecting oral medication;
4. Toxicity that is >=Grade 2 caused by previous cancer therapy;
5. Patients with congenital bleeding or coagulopathy, or are being treated with anticoagulants;
6. Patients with uncontrolled infections;
7. Has received surgery, chemotherapy, radiotherapy or other anticancer therapies 2 weeks before the first dose;
8. Has received Chinese patent medicines with anti-tumor indications that National Medical Products Administration(NMPA) approved within 2 weeks before the first dose;
9. Pleural effusion, pericardial effusion or ascites that cannot be controlled and need repeated drainage;
10. Central nervous system metastases;
11. Has participated in other clinical studies within 4 weeks before the first dose;
12. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | up to 18 months
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Maximum Tolerated Dose (MTD) | up to 18 months
  The maximum Dose at which less than 33% subjects experiencing DLT
Recommended Phase II Dose (RP2D) | up to 18 months
  RP2D will be based on evaluation of clinical safety and tolerability and guided by accumulating pharmacokinetics (PK) data
Adverse Events (AEs) | Baseline up to 24 months
  Type, frequency, seriousness and severity of adverse events and laboratory abnormalities, such as hyperuricemia.

SECONDARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) | Hour 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on single dose ; Hour 0(pre-dose) of day1, day8, day15, day22 on multiple dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on multiple dose of day28)
  Maximum plasma concentration of drug
Time to reach maximum(peak )plasma concentration following drug administration (Tmax) | Hour 0(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on single dose ; Hour 0(pre-dose) of day1, day8, day15, day22 on multiple dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on multiple dose of day28)
  Time to Maximum plasma concentration of drug
Elimination half-life (t1/2) | Hour 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on single dose ; Hour 0 (pre-dose) of day1, day8, day15, day22 on multiple dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on multiple dose of day28)
  Terminal-phase elimination half life
Overall response rate (ORR) | Baseline up to 24 months
  The sum of percentage of participants with stringent complete response rate, complete response rate, very good partial response, partial response rate in MM The sum of percentage of participants with complete response rate, partial response rate for B-NHL
Clinical benefit rate (CBR) | Baseline up to 24 months
  The sum of percentage of participants with stringent complete response rate, complete response rate, very good partial response, partial response rate, minimal response rate in MM
Time to response (TTR) | Baseline up to 24 months
  Time from the first date of dose to the first date of documented response (partial response [PR] or greater).
Duration of Response (DOR) | Baseline up to 24 months
  Time from the first documentation of response (PR or greater) to the first documentation of Progressive disease (PD) or death from any cause, whichever occurs first
Progression-free survival (PFS) | Baseline up to 24 months
  Time from the first dose to the first documentation of PD or death from any cause, whichever occurs first
Overall survival (OS) | Baseline up to 24 months
  Time from the first dose to death due to any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality